CLINICAL TRIAL: NCT04392609
Title: Predicting Locally Advanced Rectal Cancer Response to NCT and NCRT With MRI, and Comparison of MR Imaging Evaluation Between NCT and NCRT
Brief Title: Predicting Locally Advanced Rectal Cancer Response to NCT and NCRT With MRI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ziqiang Wang,MD (Other)
Responsible Party: Sponsor-Investigator, Ziqiang Wang,MD, physician, West China Hospital
Organization: West China Hospital (Other)
Other Study IDs: MR-NT-2020
Record Dates: First submitted 2020-05-10; First posted 2020-05-19 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Rectal Cancer; MRI
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This trial was designed to to study whether there is a difference in MRI image evaluation between NCRT and NCT, and try to build a model to predict the efficacy of neoadjuvant therapy by combining multiple imaging indexes.

DETAILED DESCRIPTION:
This study was designed as a retrospective case-control study. All 116 patients with locally advanced rectal cancer who started neoadjuvant chemoradiotherapy and underwent radical surgery in West of China Hospital and completed the required MR examination before and after neoadjuvant treatment were included from March 2016 to December 2019. MRI imaging indicators of patients before and after neoadjuvant therapy, including tumor location, longitudinal diameter, circumferential Angle, DWI signal, mrTRG and texture feature data, were retrospectively collected to analyze the changes before and after treatment, and compared with patients receiving NCT in PART1. At the same time, indicators with statistical differences will be included in the construction of models predicting different pathological outcomes after NCT and NCRT, and the efficacy of the models was evaluated through c-index values and ROC analysis of bootstrap resampling 500 times.

ELIGIBILITY:
Inclusion Criteria:

1. pathological diagnosis of rectal cancer;
2. received neoadjuvant chemoradiotherapy before surgery;
3. before neoadjuvant therapy and before surgery, the patients received thin and high resolution MRI examination of the rectum.
4. before neoadjuvant therapy, colonoscopy, rectal contrast-enhanced ultrasound or MRI showed that the lower margin of the tumor was within 12cm from the anal margin;
5. pre-neoadjuvant clinical stage II/III (AJCC 7th edition);

Exclusion Criteria:

1. simultaneous distant metastatic tumor should be considered at the first diagnosis;
2. patients with distant metastasis were not considered at the initial diagnosis;
3. with other malignant tumors;
4. before neoadjuvant therapy, patients had received other relevant treatments;
5. to undergo palliative surgery or emergency surgery in the course of neoadjuvant therapy;

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with locally advanced rectal cancer who started neoadjuvant chemoradiotherapy and underwent radical surgery in West of China Hospital and completed the required MR examination before and after neoadjuvant treatment were included from March 2016 to December 2019.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2020-01-15 (Actual); Primary Completion 2020-06-15 (Estimated); Study Completion 2020-07-15 (Estimated)

PRIMARY OUTCOMES:
pTRG | within 2 week after surgery
  pathological tumour regression grading

CONTACTS AND LOCATIONS:
Locations (1):
- Guoxue Road 37#,West China Hospital, Chengdu, Sichuan, China